CLINICAL TRIAL: NCT02451241
Title: The Role of Acupuncture for the Treatment of Obstructive Sleep Apnea in Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Rodrigo Pinto Pedrosa, MD, PhD, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sleep01
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Acupuncture
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- sham acupuncture (Sham Comparator): group will be submitted to placebo electroacupuncture for 20 minutes, two times a week for 5 weeks. Each session lasts about 40 min.
  Interventions: Other: acupuncture
- acupuncture (Experimental): group will be submitted to electroacupuncture for 20 minutes, two times a week for 5 weeks. Each session lasts about 40 min.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — electroacupuncture

SUMMARY:
Recent evidences from small studies show potential benefit of acupuncture in the treatment of obstructive sleep apnea (OSA). These studies did not evaluate the benefit of the treatment on the cardiovascular system.

Primary end-point:

To investigate the effects of acupuncture in improving OSA severity among hypertensive patients.

Secondary end-point To investigate the effect of acupuncture in improving the quality of life and sleep assessed by the Short Form 36 (SF-36) questionnaire and Pittsburgh Questionaire (PSQI); To investigate the effect of acupuncture in blood pressure and arterial stiffness

ELIGIBILITY:
Inclusion Criteria:

* 5<apnea-hypopnea index (AHI)<30 e/h

Exclusion Criteria:

* body mass index > 35 kg/m2
* Previous OSA treatment

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 5 weeks
  reduction in AHI

SECONDARY OUTCOMES:
Sleep quality | 5 weeks
  Improvement in PSQI scores
Pulse Wave Velocity (PWV) | 5 weeks
  reduction in PWV
Blood pressure | 5 weeks
  ambulatory blood pressure monitoring (ABPM) 24h reduction
Quality of life | 5 weeks
  Short Form 36 Health Survey (SF36) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Rodrigo Pedrosa, Recife, Pernambuco, Brazil